CLINICAL TRIAL: NCT02683564
Title: A Study of BOW015 (Infliximab-EPIRUS) and Infliximab in Patients With Active Rheumatoid Arthritis on Stable Methotrexate: The UNIFORM Study
Brief Title: BOW015 (Infliximab-EPIRUS) and Infliximab in Patients With Active Rheumatoid Arthritis: The UNIFORM Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Epirus Biopharmaceuticals (Switzerland) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPI-BOW015-003
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOW015 (Experimental): Infliximab-EPIRUS, 3mg/kg body weight as intra venous infusion at weeks 0, 2, 6 then every 8 weeks thereafter up to Week 46.
  Interventions: Drug: BOW015
- Remicade (Active Comparator): Remicade (infliximab) , 3mg/kg body weight as intra venous infusion at weeks 0, 2, 6 then every 8 weeks thereafter up to Week 46.
  Interventions: Drug: Remicade

INTERVENTIONS:
Drug: BOW015 — monoclonal antibody against TNF-alpha
  Other Names: infliximab-EPIRUS
  Arms: BOW015
Drug: Remicade — monoclonal antibody against TNF-alpha
  Other Names: infliximab
  Arms: Remicade

SUMMARY:
This is a prospective, randomized, double-blind, parallel group, multicentre global phase 3 clinical study to evaluate the efficacy, safety and immunogenicity of BOW015 (infliximab-EPIRUS) compared to Remicade in subjects with active Rheumatoid Arthritis (RA) despite Methotrexate (MTX) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female, aged 18 to 80
2. Diagnosis of Rheumatoid Arthritis (RA) according to the revised ACR/ EULAR 2010 classification criteria for RA
3. Patients must have ACR/EULAR 2010 classification criteria score ≥ 6
4. Patients must have active disease
5. Patients must have been on treatment with methotrexate

Key Exclusion Criteria:

1. Prior use of infliximab, adalimumab, certolizumab, golimumab, tocilizumab, rituximab, or etanercept or any other biological treatment
2. Patients with any prior or current use of anakinra and abatacept
3. Patients with suspected or confirmed current active tuberculosis (TB)
4. Patients with latent tuberculosis must start treatment for latent tuberculosis
5. Patients who have a current or past history of chronic infection with Hepatitis B, Hepatitis C, or infection with Human Immunodeficiency Virus-1 or-2
6. History of completely excised and cured squamous carcinoma of the uterine cervix, cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma
7. History of lymphoproliferative disease
8. History or presence of any other form of malignancy
9. Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease
10. History of congestive heart failure or unstable angina
11. History of any autoimmune disease other than RA
12. Major surgery within 12 weeks and planned major surgery
13. History of serious infection
14. Pre-existing central nervous system demyelinating disorders
15. Administration of live or live-attenuated vaccine within 4 weeks of screening
16. Clinically significant adverse reaction to murine or chimeric proteins
17. History or presence of any medical or psychiatric condition or disease, or clinically significant laboratory abnormality
18. Participation in any clinical study of an investigational product within the previous 3 months prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR) 20 clinical response | 16 weeks

SECONDARY OUTCOMES:
ACR20 | 54 weeks
Diseases Activity Score (DAS)28 calculated with C-reactive protein (CRP) | 54 weeks
Health Assessment Questionnaire-Disability Index (HAQ-DI) | 54 weeks